CLINICAL TRIAL: NCT06176105
Title: Mortality After Transfusion of Ever-pregnant Donor Red Blood Cells
Acronym: MATER
Status: Completed | Type: Observational
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Responsible Party: Sponsor
Other Study IDs: PPOC 18-03
Record Dates: First submitted 2023-11-22; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2019-03

CONDITIONS: Anemia
Keywords: Transfusion; Red blood cells; Sex mismatch; Pregnancy
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The MATER study is an observational cohort study on first ever transfusion recipients in six hospitals in the Netherlands, with information collected on both donor and patient characteristics. We aim to further specify which combination of characteristics of both donors and patients determine the increased risk of mortality after blood transfusions.

DETAILED DESCRIPTION:
Background In 2011, a link between donor sex and death of transfusion recipients was observed in red blood cell transfusions (Middelburg et al., Vox Sanquinis, 2011). This was further investigated by Caram-Deelder et al., who showed the transfusion of red blood cells from ever-pregnant donors was associated with higher mortality in young men (with age up to 50 years) (Caram-Deelder et al., JAMA, 2017). However, the biological mechanisms explaining this association remained unclear. More data is needed to be able to specify which combination of characteristics of both donors and patients determines this increased risk of mortality after red blood cell transfusions. Therefore, the MATER study was initiated: 'Mortality After Transfusion of Ever-pregnant donor Red blood cells'. Here, we aim to validate previous research on the association between donor pregnancy history and transfusion recipient mortality.

Rationale Red blood cells constitute the biggest part of the blood supply. They are currently transfused without consideration of the sex of the blood donor and the recipient. Recent evidence shows such a policy to be associated with increased mortality in male recipients of red blood cells from female donors with a history of pregnancy. This project aims to find clues for the biological mechanism behind this association. This knowledge will allow for more personalized future transfusion strategies that will minimize both side effects and associated mortality of recipients of red blood cell transfusions.

Methodology First-ever transfusion recipients in the Netherlands between 2005 and 2018 which were performed in the hospitals participating in the R-FACT study will be included in this study. All blood donations and the corresponding donors linked to these recipients will be included in this study. Cox regression analysis will be used to assess the effect of donor pregnancy on transfusion recipient mortality. This analysis method allows modelling the relation between exposure (donor pregnancy history), outcome (mortality), and confounders (e.g. total number of transfusions, year of transfusion, ABO and Rh blood type, sex of the patient, and hospital) taking into account that exposure and confounders vary over time. Pregnancy history will be investigated as number of pregnancies, time since last pregnancy, different partners and type of pregnancy (i.e. boy versus girl pregnancies, outcome of pregnancy). The hazard ratio will be presented for exposure to blood products with different characteristics, stratified by patient age, sex and (if possible) transfusion indication. Effect modification by storage time will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* have received a first transfusion between 20-03-2004 and 31-12-2018 in one of the hospitals participating in the R-FACT study OR
* have donated blood for a blood product which was used in one of the hospitals participating in the R-FACT study between 20-03-2004 and 31-12-2018

Exclusion Criteria:

* N.A.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First ever red blood cell transfusion recipients in the Netherlands between 20-03-2004 and 31-12-2018 which were performed in the hospitals participating in the R-FACT study will be included in this study. All blood donations and the corresponding donors linked to these recipients will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 101000 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 2015-2018
  In total, this cohort contains data on over 100,000 first-ever transfusion recipients and their received transfusions from six hospitals in the Netherlands, with information collected on both donor and patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: J van der Bom, Prof, Principal Investigator — Jon J van Rood Center for Clinical Transfusion Research
Locations (1):
- Sanquin blood bank, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caram-Deelder C, Kreuger AL, Evers D, de Vooght KMK, van de Kerkhof D, Visser O, Pequeriaux NCV, Hudig F, Zwaginga JJ, van der Bom JG, Middelburg RA. Association of Blood Transfusion From Female Donors With and Without a History of Pregnancy With Mortality Among Male and Female Transfusion Recipients. JAMA. 2017 Oct 17;318(15):1471-1478. doi: 10.1001/jama.2017.14825. PMID 29049654
- [Background] Middelburg RA, Briet E, van der Bom JG. Mortality after transfusions, relation to donor sex. Vox Sang. 2011 Oct;101(3):221-9. doi: 10.1111/j.1423-0410.2011.01487.x. Epub 2011 Apr 8. PMID 21477152